CLINICAL TRIAL: NCT07144319
Title: Exploration of Novel AI-enabled Blue Light Enhanced Cystoscopy
Acronym: ENAiBLE
Status: Not yet recruiting | Type: Observational
Sponsor: Photocure (Industry)
Responsible Party: Sponsor
Other Study IDs: PCAIX01/25
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Bladder Cancer; Non-muscle Invasive Bladder Cancer
Keywords: bladder cancer; artificial intelligence; cystoscopy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BLC patients: Adult, consenting patients scheduled for BLC as part of clinical practice.

SUMMARY:
Blue light cystoscopy (BLC) is a diagnostic procedure in bladder cancer where the inside of the bladder is observed with a camera to detect bladder lesions. Unlike regular white light cystoscopy, blue light cystoscopy makes use of a drug that induces fluorescence under blue light preferentially in neoplastic and malignant cells that helps visualize bladder lesions during the cystoscopic procedure. Blue light cystoscopy has shown to improve detection of bladder cancer.

Cystoscopy, including blue light cystoscopy, is a procedure involving assessment of the visual appearance of the bladder surface, leading to decisions of taking biopsies, remove suspicious areas and assign treatment options. The assessment is subjective and has a large operator variability. These shortcomings show an opportunity for computer aided detection (CADe) medical device to add value to both clinicians and patients.

The objective of this data collection study is to build a high-quality, diverse data set of video, image recordings and relevant clinical data from BLC procedures performed as part of routine clinical practice to train a computer-aided detection (CADe) algorithm for real- time lesion detection during cystoscopy. The data will be used to support the training, non-clinical technical development and testing of such AI algorithms for use during cystoscopy and to provide documentation needed for training of such algorithms and to assist in guiding future validation of such algorithms.

Exploratory purposes of the study is to use data to explore future AI algorithms in bladder cancer, such as computer-aided diagnosis (CADx) AI algorithms, image enhancement and cystoscopy improvement algorithms, including bladder mapping, tumor visualization, cystoscopy documentation, and combination models of image and clinical data including risk assessment, clinical outcomes, and disease modeling

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Written informed consent, approved by relevant IRB/IEC, signed
* Hexvix/Cysview has been prescribed in the usual manner in accordance with the terms of the marketing authorization (see Appendix B)
* Physician has planned to do a blue light cystoscopy on the patient and to obtain biopsies, if clinically indicated, of suspicious lesions with video confirmation.
* Patient has not previously taken part in this study

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Routine clinical practice patients scheduled for BLC
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Video and image collection | 1 day
  To collect videos, images and relevant clinical data from BLC procedures performed as part of clinical practice. The data will be used to explore the potential of a BLC-enabled AI algorithm for lesion detection of bladder cancer.

IPD SHARING:
Plan to Share IPD: No